CLINICAL TRIAL: NCT05387447
Title: The Loneliness Epidemic Tailoring Interventions to Reduce Loneliness and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0177-21-EP
Record Dates: First submitted 2022-05-12; First posted 2022-05-24 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pain, Chronic; Loneliness
Keywords: Older Adults; Pain; Loneliness; Voice Assistant Technology
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conversational Voice Assistant (Enhanced) (Experimental): Participants will complete a personalized and tailored interactive routine with the voice assistant.
  Interventions: Behavioral: Conversational Voice Assistant (Standard)
- Conversational Voice Assistant (Standard) (Experimental): Participants will complete a standard interactive routine with the voice assistant.
  Interventions: Behavioral: Conversational Voice Assistant (Enhanced)

INTERVENTIONS:
Behavioral: Conversational Voice Assistant (Enhanced) — Interactive routine is based on tailoring to the participants type of pain and personality.
  Arms: Conversational Voice Assistant (Standard)
Behavioral: Conversational Voice Assistant (Standard) — Interactive routine is a basic interaction with the voice assistant.
  Arms: Conversational Voice Assistant (Enhanced)

SUMMARY:
Approximately 24% of community-dwelling older adults are socially isolated, and over 40% of adults 60 and older report feeling lonely. Over 50% of midlife and older adults who perceive their health as fair or poor are lonely in contrast to 27% percent who believe their health to be excellent or very good. Loneliness has been associated with high mortality and inflammation which can influence symptoms such as pain. Social isolation and pain further contribute to loneliness. Studies have reported one and a half greater odds of being socially isolated among older adults with clinical osteoarthritis (OA) of the hip and/or knee than someone with similar characteristics without OA. Pain is significant because it is highly prevalent among older adults and is associated with disability, social isolation, and greater costs and burden to health care systems. A recent review of the literature found that several interventions influence social isolation and loneliness. As these interventions require in-person interaction, those who are socially isolated or distanced due to pain may not benefit due to a lack of access. Current advancements in technology and social media may provide opportunities to reduce loneliness and pain due to social isolation. Online and technology-based interventions have shown potential to engage older adults to improve communication and social connection. Given that socialization with these approaches are supportive only when the other person is available for that interaction. An intervention that utilizes technology to incorporate solitary interventions may be efficacious. Studies found a trend for a positive relationship between the use of a voice assistant and loneliness in aging adults living alone.

Building upon this evidence on loneliness and pain research, conversational voice assistant (CVA) technology and personalized persuasion, investigators will conduct a 12-week randomized control pilot with older adults that live alone and self-report pain. Participants will interact with a standard or a personally enhanced loneliness routine delivered through a CVA. Investigators will explore intervention feasibility and examine the efficacy of both standard and personalized interventions on loneliness and secondary outcomes.

DETAILED DESCRIPTION:
Approximately 24% of community-dwelling older adults are socially isolated, and over 40% of adults 60 and older report feeling lonely. Over 50% of midlife and older adults who perceive their health as fair or poor are lonely in contrast to 27% percent who believe their health to be excellent or very good. Loneliness has been associated with high mortality and inflammation which can influence symptoms such as pain. Social isolation and pain further contribute to loneliness. Studies have reported one and a half greater odds of being socially isolated among older adults with clinical osteoarthritis (OA) of the hip and/or knee than someone with similar characteristics without OA. Pain is significant because it is highly prevalent among older adults and is associated with disability, social isolation, and greater costs and burden to health care systems. A recent review of the literature found that several interventions influence social isolation and loneliness. As these interventions require in-person interaction, those who are socially isolated or distanced due to pain may not benefit due to a lack of access. Current advancements in technology and social media may provide opportunities to reduce loneliness and pain due to social isolation. Online and technology-based interventions have shown potential to engage older adults to improve communication and social connection. Given that socialization with these approaches are supportive only when the other person is available for that interaction. An intervention that utilizes technology to incorporate solitary interventions may be efficacious. Studies found a trend for a positive relationship between the use of a voice assistant and loneliness in aging adults living alone.

Investigators propose to conduct a 12-week pilot trial with participants randomly assigned to either the conversational voice assistant-standard group (CVA-S) or the conversational voice assistant-enhanced loneliness routine treatment group (CVA-ELR). Data will be collected at pre- (baseline) and post-intervention (after 12-weeks). The 12-week duration was chosen based on published intervention studies designed to reduce loneliness in older adults. Both groups will receive basic training on how to use the conversational voice assistant.

The CVA-S group will receive an a priori set of evidence-based interactions to perform with the conversational voice assistant. The interaction will be 15 minutes, performed once in the morning and once in the evening, at preset times. The participants will do a meditation activity, play an interactive trivia game, and ask the assistant to tell a joke. These activities were selected based on prior literature. The CVA-ELR group will receive personalized intervention materials based on individual baseline personality and entertainment inventory results. Potential personalization tactics used to match intervention materials with each individual's personality and entertainment preferences include identification (name integration), expectation (customization claim), contextualization (meaningful personal context), descriptive (personal data), comparative (contrast to others), evaluative (personal recommendation). Both interventions will use the minimum viable user experience (UX) design approach to develop intervention materials and will be delivered through a smart speaker. Investigator developed questionnaires will be used to collect self-reported descriptive demographic and health history.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years of age
* Live alone (single-family home, independent, or assisted living)
* Experienced or currently experiencing musculoskeletal pain
* Wireless internet access via a broadband Internet connection

Exclusion Criteria:

* Memory loss as evidenced by poor performance on the Mini Cog (0 to 2 points)
* Inability to speak English
* Prior or current use of a conversational voice assistant
* Unwilling to engage with the voice assistant

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Y Shade, PhD, RN, Principal Investigator — University of Nebraska
Locations (4):
- United States (4):
  - The Legacy, Lincoln, Nebraska
  - Eastmont Senior Living Apartments, Lincoln, Nebraska
  - Trinity Courtyard, Omaha, Nebraska
  - Aksarben Village Senior Apartments, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from Aksarben Village Senior Apartments, Trinity Courtyard Senior Apartments, Eastmont Senior Living Apartments, The Legacy Senior Living apartments
Groups:
- Conversational Voice Assistant-Standard: Participants will complete a standard interactive routine with the voice assistant.
  Conversational Voice Assistant-Standard: Interactive routine is a basic interaction with the voice assistant.
- Conversational Voice Assistant-Enhanced: Participants will complete a personalized and tailored interactive routine with the voice assistant.
  Conversational Voice Assistant-Enhanced: Interactive routine is based on tailoring to the participants type of pain and personality.
Period: Overall Study
Arm/Group | Conversational Voice Assistant-Standard | Conversational Voice Assistant-Enhanced
Started | 28 | 30
Completed | 25 | 25
Not Completed | 3 | 5
Not completed — Participants changed their minds about study participation. | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conversational Voice Assistant-Standard | Conversational Voice Assistant-Enhanced | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.32 (7.83) | 78.9 (7.76) | 79 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 51
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 28 | 29 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 30 | 58
Self-reported Pain Severity [Mean (Full Range); unit: units on a scale] — Self-reported pain severity will be recorded using the Brief Pain Inventory Short Form. Scores range from 0 as minimal score meaning no pain or pain interference to 10 as maximum score that equates to severe pain or complete pain interference. Higher scores indicate worse symptoms.
  units on a scale
    Pain Severity | 3.42 [0 to 9.5] | 3.76 [0 to 7.5] | 3.6 [0 to 9.5]
    Pain Interference | 3.66 [0 to 8] | 4.56 [1.29 to 7.43] | 4.12 [0 to 8]
Self-Reported Loneliness [Mean (Full Range); unit: units on a scale] — Self-reported loneliness will be recorded using the University of California Los Angeles Loneliness Scale. The range of scores is 20 minimum to 80 as the maximum. The cut-offs for loneliness severity: <28 = no/low loneliness, 28 to 43 = moderate loneliness, and total score >43 = high loneliness. Higher scores indicate worse self-reported loneliness. Scores will be compared between groups at baseline and 12-weeks post-intervention.
  units on a scale | 62.27 [40 to 79] | 67.78 [45 to 78] | 65.14 [40 to 79]
Geriatric Depression [Mean (Full Range); unit: units on a scale] — Self-reported depressive symptoms will be recorded. Scores range from 0 as a minimum to a 15 as a maximum. Higher scores indicate worse depression: 0-4 normal, 5-8 mild depression, 9-11 moderate depression, and 12-15: severe depression. Scores will be compared between groups at baseline and 12-weeks post-intervention.
  units on a scale | 6.92 [4 to 11] | 7.79 [4 to 12] | 7.10 [4 to 12]
Self-efficacy for Managing Symptoms [Mean (Full Range); unit: units on a scale] — Self-reported self-efficacy or confidence in managing pain symptoms will be recorded using Patient-Reported Outcomes Measurement Information System (PROMIS). Scores range from a minimum of 0 to a maximum of 100. A score of 50 represents the average. Higher scores above 50 indicate better self-reported self-efficacy in managing pain. Scores will be compared between groups at baseline and 12-weeks post-intervention.
  units on a scale | 34 [26 to 40] | 32 [19 to 40] | 33 [19 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Pain Severity
Description: Self-reported pain severity will be recorded using the Brief Pain Inventory Short Form. Scores range from 0 as minimal score meaning no pain or pain interference to 10 as maximum score that equates to severe pain or complete pain interference. Higher scores indicate worse symptoms.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Conversational Voice Assistant (Standard): Participants will complete a standard interactive routine with the voice assistant.
  Conversational Voice Assistant-Standard: Interactive routine is a basic interaction with the voice assistant.
- Conversational Voice Assistant (Enhanced): Participants will complete a personalized and tailored interactive routine with the voice assistant.
  Conversational Voice Assistant-Enhanced: Interactive routine is based on tailoring to the participants type of pain and personality.
Arm/Group | Conversational Voice Assistant (Standard) | Conversational Voice Assistant (Enhanced)
Number analyzed (Participants) | 25 | 25
score on a scale
  Brief Pain Inventory Pain Interference | 2.57 (2.11) | 3.71 (2.36)
  Brief Pain Inventory Pain Severity | 3.22 (2.21) | 3.89 (2.69)
Statistical Analysis 1: Comparison: Conversational Voice Assistant (Standard) vs Conversational Voice Assistant (Enhanced); Test type: Other; p = .05, Z score

2. Primary Outcome: Self-reported Loneliness
Description: Self-reported loneliness will be recorded using the University of California Los Angeles Loneliness Scale. The range of scores is 20 minimum to 80 as the maximum. The cut-offs for loneliness severity: <28 = no/low loneliness, 28 to 43 = moderate loneliness, and total score >43 = high loneliness. Higher scores indicate worse self-reported loneliness. Scores will be compared between groups at baseline and 12-weeks post-intervention.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conversational Voice Assistant-Standard | Conversational Voice Assistant-Enhanced
Number analyzed (Participants) | 25 | 25
score on a scale | 58.83 (19.73) | 58.84 (15.95)
Statistical Analysis 1: Comparison: Conversational Voice Assistant-Standard vs Conversational Voice Assistant-Enhanced; Test type: Other; p = .05, Z score

3. Secondary Outcome: Conversational Voice Assistant System Usability
Description: Self-reported ease of use of the voice assistant routines will be recorded. Score range from a minimum of 0 and a maximum of 100. Higher scores mean better usability: 0-51 "awful" or "poor" usability (significant problems), 51-68 "okay" usability (room for improvement), 68-80.3 "good" usability, 80.3+ "excellent" usability (highly usable system). Scores will be compared between groups at 12-weeks post-intervention.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Conversational Voice Assistant (Standard): Participants will complete a basic (standard) interactive routine with the Conversational Voice Assistant.
- Conversational Voice Assistant (Enhanced): Participants will complete a personalized interactive routine with the Conversational Voice Assistant that is tailored to the participants type of pain and personality.
Arm/Group | Conversational Voice Assistant (Standard) | Conversational Voice Assistant (Enhanced)
Number analyzed (Participants) | 25 | 25
score on a scale | 66.29 (6.94) | 74.5 (11.9)

4. Secondary Outcome: Geriatric Depression
Description: Self-reported depressive symptoms will be recorded. Scores range from 0 as a minimum to a 15 as a maximum. Higher scores indicate worse depression: 0-4 normal, 5-8 5ild depression, 9-11 moderate depression, and 12-15: severe depression. Scores will be compared between groups at baseline and 12-weeks post-intervention.
Time Frame: Baseline and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conversational Voice Assistant-Standard | Conversational Voice Assistant-Enhanced
Number analyzed (Participants) | 25 | 25
score on a scale | 6.25 (2.36) | 6.65 (2.54)
Statistical Analysis 1: Comparison: Conversational Voice Assistant-Standard vs Conversational Voice Assistant-Enhanced; Test type: Other; p = .05, Z score

5. Secondary Outcome: Self-efficacy for Managing Symptoms
Description: Self-reported self-efficacy or confidence in managing pain symptoms will be recorded using Patient-Reported Outcomes Measurement Information System (PROMIS). Scores range from a minimum of 0 to a maximum of 100. A score of 50 represents the average. Higher scores above 50 indicate better self-reported self-efficacy in managing pain. Scores will be compared between groups at baseline and 12-weeks post-intervention.
Time Frame: Baseline and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conversational Voice Assistant-Standard | Conversational Voice Assistant-Enhanced
Number analyzed (Participants) | 25 | 25
score on a scale | 34 (7.56) | 31 (8.41)
Statistical Analysis 1: Comparison: Conversational Voice Assistant-Standard vs Conversational Voice Assistant-Enhanced; Test type: Other; p = .05, Z score

ADVERSE EVENTS:
Time Frame: Every two weeks post enrollment for 3 months.
Arm/Group | Conversational Voice Assistant-Standard | Conversational Voice Assistant-Enhanced
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Those without regular internet access in their home due to location (e.g. rural areas) or lack of broadband access (due to personal choice or financial restraints) would not be able to interact with conversational voice assistants. Our participants self-reported pain and loneliness, but our study may not have enrolled individuals who are on the highest extremes of experiencing symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT05387447/Prot_SAP_000.pdf